CLINICAL TRIAL: NCT00926406
Title: Environmental Exposure to Lead and Its Health Effects on Patients With Maintenance Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Institutional Review Board, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 96-1455C
Record Dates: First submitted 2009-06-21; First posted 2009-06-23 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Malnutrition; Inflammation; Lead Poisoning
Keywords: Environmental lead exposure, maintenance hemodialysis; blood lead levels, EDTA chelating agents, malnutrition, anemia, inflammation, mortality.; To determine whether lead chelation therapy improves the anemia, malnutrition, inflammation, morbidity or mortality in hemodialysis patients.
MeSH Terms: conditions — Anemia; Malnutrition; Inflammation; Lead Poisoning

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: lead chelation therapy — Patients with lead poisoning (BLL> 20μg/dl) are randomly assigned to a control or chelation group, on the 1:1 proportion. During the 3 months, 50 chelation group patients receive 2-hour weekly intravenous infusions of one vial (1 g) of calcium di-sodium EDTA mixed with 200 ml of normal saline until BLB is BLL < 5 μg/dl. Fifty control patients receive weekly 2-hour infusions of one vial (20 ml) of 50% glucose mixed with 200 ml of normal saline over a period of 12 weeks9.

SUMMARY:
One thousand patients with LHD who have no history of exposure to lead will be observed for 18 months. Blood lead level(BLL), biochemical data, hemoglobin, albumin, Cr, high sensitivity C-reactive protein (HsCRP), and blood cell counts are assessed at baseline. The morbidity and mortality are recorded in detail. Then, one hundred subjects with high BLL (>20μg/dl) will be randomly assigned to the study and control groups. For 3-6 months, the 50 patients in the study group will receive lead-chelation therapy with calcium disodium EDTA weekly until the BLB falls below BLL< 5 μg/dl, and the 50 control group patients receive weekly placebo for 12 weeks. During the ensuing 18 months, the BLL, biochemical data will be regularly followed up every 3 months. BLL is measured every 6 months. If BLL of the study group patients increase >10 μg/dl, the chelation therapy will be performed again until their BLL is <5 μg/dl. The primary end point is morbidity or mortality during the observation and follow-up period. A secondary end point is the change in hemoglobin, albumin, Cr and Hs CRP during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* MHD patients have dialyzed for more than 6 months and age >18 and < 90 year-old

Exclusion Criteria:

* Patients with malignancies and obvious infectious diseases as well as those who are hospitalized or underwent surgery or renal transplantation within the 3 months preceding the investigation;Patients with a history of occupational exposure to heavy metals, metal intoxication, living in metal-contaminated areas were also excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point is morbidity or mortality during the follow-up period. | 18 months follow-up period

SECONDARY OUTCOMES:
A secondary end point is the change in HB, albumin, Cr and Hs CRP during the follow up period. | 18 months follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan